CLINICAL TRIAL: NCT00806676
Title: Antibody Response to Human Papillomavirus Recombinant Vaccine (Gardasil®) in Girls and Young Women With Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NA_00020699
Record Dates: First submitted 2008-12-09; First posted 2008-12-11 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; children; dialysis; kidney transplant; human papilloma virus; Gardasil; Chronic kidney disease (non-dialysis, dialysis, and kidney transplant) secondary to any cause.
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1. Chronic Kidney Disease, NKF Stage 1-4 (Other): Gardasil vaccine series will be administered according to FDA-approved schedule, as recommended by the Centers for Disease Control and Prevention and the American Academy of Pediatrics. Geometric antibody titers among those with chronic kidney disease will be compared to titers in the general population measured during Phase III clinical studies by Merck & Co, Inc, to prove efficacy of the vaccine and obtain FDA approval.
  Interventions: Drug: Gardasil® Vaccine (FDA-approved vaccination regimen)
- 2. ESRD (dialysis) (Other): Gardasil vaccine series will be administered according to FDA-approved schedule, as recommended by the Centers for Disease Control and Prevention and the American Academy of Pediatrics. Geometric antibody titers among those with ESRD will be compared to titers in the general population measured during Phase III clinical studies by Merck & Co, Inc, to prove efficacy of the vaccine and obtain FDA approval.
  Interventions: Drug: Gardasil® Vaccine (FDA-approved vaccination regimen)
- 3. Kidney Transplant Recipient (Other): Gardasil vaccine series will be administered according to FDA-approved schedule, as recommended by the Centers for Disease Control and Prevention and the American Academy of Pediatrics. Geometric antibody titers among those with a kidney transplant will be compared to titers in the general population measured during Phase III clinical studies by Merck & Co, Inc, to prove efficacy of the vaccine and obtain FDA approval.
  Interventions: Drug: Gardasil® Vaccine (FDA-approved vaccination regimen)

INTERVENTIONS:
Drug: Gardasil® Vaccine (FDA-approved vaccination regimen) — Standard Gardasil® 3-dose regimen (0.5 mL/dose; doses at 0, 2 and 6 months) delivered to females with chronic kidney disease 9-21 years of age.

SUMMARY:
People with chronic kidney disease are known to have immune response abnormalities, including a diminished response to some vaccinations. Those with chronic kidney disease have a disproportionate burden of HPV 6-, 11-, 16- and/or 18-related genital tract disease. Due to immune response abnormalities, the CKD population may or may not respond to the recommended three-dose regimen of Gardasil®, a vaccine intended to protect against HPV 6-, 11-, 16-, and 18-related genital tract disease. The objective of this study is to measure the antibody response to Gardasil® in female patients 9-21 years of age with chronic kidney disease (CKD) (Stage 1-4), end-stage kidney disease (Stage 5 CKD), and status-post kidney transplant. Gardasil® vaccine will be administered according to the FDA-approved schedule. Blood samples to measure antibody levels to vaccine strains of human papillomavirus (HPV) will be obtained at months 0, 7 and 24.

ELIGIBILITY:
Inclusion Criteria:

Females, aged 9-21 years, in the following groups:

* CKD (defined as estimated glomerular filtration rate between 90 ml/min/1.73m2 and 15 ml/min/1.73m2, as calculated by the Schwartz formula)
* ESRD (eGFR < 15 ml/min/1.73m2, or receiving chronic dialysis [peritoneal or hemodialysis])
* Status-post kidney transplant

Exclusion Criteria:

* Within first 3 months post kidney transplant
* Within 3 months of kidney rejection episode
* Hypersensitivity to active substances or excipients of Gardasil vaccine

Ages: 9 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 67 (Actual)
Dates: Start 2008-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Fadrowski, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Emory Healthcare & Children's Healthcare of Atlanta Pediatric Nephrology Clinic, Atlanta, Georgia
  - Johns Hopkins University Harriet Lane Kidney Center, Rubenstein Child Health Bldg, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1. Chronic Kidney Disease, NKF Stage 1-4 | 2. ESRD (Dialysis) | 3. Kidney Transplant Recipient
Started | 29 | 9 | 29
Completed | 25 | 9 | 23
Not Completed | 4 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1. Chronic Kidney Disease, NKF Stage 1-4 | 2. ESRD (Dialysis) | 3. Kidney Transplant Recipient | Total
Number analyzed (Participants) | 25 | 9 | 23 | 57
Age, Customized [Count of Participants; unit: Participants]
  >=11, <=21, years | 25 | 9 | 23 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 9 | 23 | 57
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 4 | 6 | 20
  White | 12 | 2 | 14 | 28
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients 9-15 Years of Age With CKD Achieving Seropositivity (IgG Assay) at Blood Draw 2
Description: The primary outcome was antibody response to each of four HPV genotypes contained within the HPV vaccine at the time periods specified for the blood draws. Antibody levels, measured by Merck GmbH, were initially determined using the competitive Luminex immunoassay(cLIA; Merck GmbH), the assay used in the original licensing studies. Seropositivity was defined as being above thresholds set at 20, 16, 20, and 24 milliMerck units for HPV genotypes 6, 11, 16, and 18, respectively, as determined in phase 2 studies among patients who were immunocompetent. Antibody levels were reanalyzed using the newer, more sensitive IgG cLIA in stored serum from blood draws 2 and 3. Seropositivity for this assay was defined as being above thresholds set at 15, 15, 7, and 10 milliMerck units for HPV genotypes 6, 11, 16, and 18, respectively.
Time Frame: Month 7
Population: Some patients did not complete all 3 blood draws because of (1) previous vaccination at primary care physician's office, which precluded blood draws 1 and/or 2; (2) inconsistent clinic visits, which precluded the 2nd or 3rd blood draw; and/or (3) administrative censoring in July 2012.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- HPV 6: HPV genotype
Arm/Group | HPV 6 | HPV 11 | HPV 16 | HPV 18
Number analyzed (Participants) | 10 | 10 | 10 | 10
percentage of participants | 100 [69 to 100] | 100 [69 to 100] | 100 [69 to 100] | 100 [69 to 100]

2. Primary Outcome: Percentage of Patients 16-21 Years of Age With CKD Achieving Seropositivity (IgG Assay) at Blood Draw 2
Time Frame: Month 7
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HPV 6 | HPV 11 | HPV 16 | HPV 18
Number analyzed (Participants) | 8 | 8 | 8 | 8
percentage of participants | 100 [63 to 100] | 100 [63 to 100] | 100 [63 to 100] | 100 [63 to 100]

3. Primary Outcome: Percentage of Patients 9-15 Years of Age on Dialysis Achieving Seropositivity (IgG Assay) at Blood Draw 2
Time Frame: Month 7
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HPV 6 | HPV 11 | HPV 16 | HPV 18
Number analyzed (Participants) | 6 | 6 | 6 | 6
percentage of participants | 100 [54 to 100] | 100 [54 to 100] | 100 [54 to 100] | 100 [54 to 100]

4. Primary Outcome: Percentage of Patients 16-21 Years of Age on Dialysis Achieving Seropositivity (IgG Assay) at Blood Draw 2
Time Frame: Month 7
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HPV 6 | HPV 11 | HPV 16 | HPV 18
Number analyzed (Participants) | 3 | 3 | 3 | 3
percentage of participants | 100 [29 to 100] | 100 [29 to 100] | 100 [29 to 100] | 100 [29 to 100]

5. Primary Outcome: Percentage of Patients 9-15 Years of Age With a Kidney Transplant Achieving Seropositivity (IgG Assay) at Blood Draw 2
Time Frame: Month 7
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HPV 6 | HPV 11 | HPV 16 | HPV 18
Number analyzed (Participants) | 8 | 8 | 8 | 8
percentage of participants | 88 [47 to 100] | 75 [35 to 97] | 100 [63 to 100] | 88 [47 to 100]

6. Primary Outcome: Percentage of Patients 16-21 Years of Age With a Kidney Transplant Achieving Seropositivity (IgG Assay) at Blood Draw 2
Time Frame: Month 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HPV 6 | HPV 11 | HPV 16 | HPV 18
Number analyzed (Participants) | 14 | 14 | 14 | 14
percentage of participants | 50 [23 to 77] | 57 [29 to 82] | 100 [77 to 100] | 64 [35 to 87]

ADVERSE EVENTS:
Arm/Group | 1. Chronic Kidney Disease, NKF Stage 1-4 | 2. ESRD (Dialysis) | 3. Kidney Transplant Recipient
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/9 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/9 | 0/23
Other Adverse Events (participants affected / at risk) | 4/25 | 0/9 | 4/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1. Chronic Kidney Disease, NKF Stage 1-4 (N=25) | 2. ESRD (Dialysis) (N=9) | 3. Kidney Transplant Recipient (N=23)
Pain at vaccine injection site (Injury, poisoning and procedural complications) | 4 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No